CLINICAL TRIAL: NCT03273491
Title: Self-weighing's Psychological Effects: a Randomized Controlled Trial Using Ecological Momentary Assessment
Brief Title: Self-Weighing: an Ecological Momentary Assessment
Acronym: SWEMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Carly R Pacanowski, Assistant Professor (2C1001), University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17A00813
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Daily Self-weighing; Daily Temperature-taking
Keywords: self-weighing; weight gain; Ecological Momentary Assessment; mood; emerging adulthood; obesity; eating disorders
MeSH Terms: conditions — Weight Gain; Obesity; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Self-Weighing Group (Experimental): Participants will be provided with a scale and instructions necessary to engage in daily self-weighing, first thing in the morning for the next three months.
  Height and weight will be measured using standard procedures
  Questionnaires will be administered at baseline and EOT: Sociodemographic questions (i.e. age, race/ethnicity, self-weighing frequency, weight goals will be collected at baseline. To assess factors that may modify reaction to intervention condition,a questionnaire will assess participant's eating attitudes, behaviors, and perception of their body.
  Questionnaires (baseline, end of Week 1, 2, 3, 4 and EOT): In order to compare results with published studies assessing constructs over varying time frames, self-esteem, anxiety, and depression will be measured at baseline, weekly for the first month, and again at EOT.
  Interventions: Behavioral: daily self-weighing
- Daily Temperature-Taking Group (Active Comparator): Participants will be provided with a thermometer and instructions necessary to engage in daily temperature-taking, first thing in the morning for the next three months.
  Height and weight will be measured using standard procedures
  Questionnaires will be administered at baseline and EOT: Sociodemographic questions (i.e. age, race/ethnicity, self-weighing frequency, weight goals will be collected at baseline. To assess factors that may modify reaction to intervention condition,a questionnaire will assess participant's eating attitudes, behaviors, and perception of their body.
  Questionnaires (baseline, end of Week 1, 2, 3, 4 and EOT): In order to compare results with published studies assessing constructs over varying time frames, self-esteem, anxiety, and depression will be measured at baseline, weekly for the first month, and again at EOT.
  Interventions: Behavioral: daily temperature-taking

INTERVENTIONS:
Behavioral: daily self-weighing — Participants are provided with a wifi-enabled scale and asked to weigh themselves daily, first thing in the morning.
  Arms: Daily Self-Weighing Group
Behavioral: daily temperature-taking — Participants are provided with a wifi-enabled thermometer and asked to take their temperature daily, first thing in the morning.
  Arms: Daily Temperature-Taking Group

SUMMARY:
The primary objective of this study is to experimentally test the momentary and more distal psychological effects of daily self weighing as compared to an active control group.

DETAILED DESCRIPTION:
Two significant public health problems, obesity and eating disorders, are prevalent during emerging adulthood, a unique stage of life between ages 18 and 25. Over half of emerging adults experience weight gain and/or disordered eating (e.g. overly restrictive dieting, binge eating); both of which contribute to obesity. Because many emerging adults attend college, the college community represents a viable population for implementing interventions to prevent weight gain, while not triggering disordered eating.

A promising strategy for preventing weight gain during college is daily self-weighing, an example of behavioral self-monitoring, an evidence-based strategy for weight control. Self-monitoring is fundamental to behavior change: feedback allows the user to evaluate progress in relation to a goal and modify behavior. Despite self-monitoring being recommended, some evidence suggests that self-monitoring strategies, self-weighing in particular, may have unintended psychological consequences; the concern being that negative mood states could precipitate disordered eating. Alternatively, other evidence suggests positive psychological outcomes related to daily self-weighing in young adults.

Technological advances have allowed for users to track personal health information in real time. Given that 60% of U.S. adults track weight, diet, or exercise, and 92% of adults aged 18-34 own a smartphone, electronic self-monitoring is feasible in this population. What is less known is individuals' psychological and behavioral response to self-monitoring. This original, important study will contribute to the fields of obesity and eating disorders and experimentally test the psychological effects of this daily weight-control intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between the ages of 18 and 26
* UD student
* Owns a smart phone
* If participant does not currently have an eating disorder or has never had one in the past

Exclusion Criteria:

* If participant currently has an eating disorder or has had one in the past
* If participant answers "yes" to 3 or more items in SCOFF

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 55 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
psychological response to daily self-weighing | 3 Months
  1. Daily self-weighing will result in significantly greater reactivity than daily-temperature-taking
  2. There will be no significance in mood ratings between daily self-weighing and daily temperature-taking groups for EMA recordings later in the day.
  3. The daily self-weighing group will report significantly more weight control behaviors at the end of the day as compared to the daily temperature-taking group.

SECONDARY OUTCOMES:
Identify moderators of response to daily self-weighing in a college-aged female population | 3 Months
  1. Participants with lower baseline dietary restraint scores will experience significantly greater success in preventing weight gain over 3 months in response to daily self-weighing as compared to daily temperature-taking, in comparison to those with higher baseline dietary restraint scores
  2. Participants with higher baseline body satisfaction, lower body consciousness, and higher-self esteem will have significantly more favorable reactions to daily self-weighing, both in terms of momentary mood and prevention of weight gain over 3 months
  3. Baseline weight status will moderate the effectiveness of daily self-weighing as a weight gain prevention tool, such that it will work significantly better for overweight patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes